CLINICAL TRIAL: NCT01677923
Title: Phase 3: Effect of Diet, Physical Activity and Insulin Sensitizer Metformin on Obesity and Associated Risks in Children and Adolescents.
Brief Title: Obesity in Children and Adolescents: Associated Risks and Early Intervention
Acronym: OCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Rasa Verkauskiene, Professor, Head of Department and Institute of Endocrinology, Lithuanian UHS, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE-2-1
Record Dates: First submitted 2012-07-30; First posted 2012-09-03 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: weight; body mass index; lipid profile; glucose profile
MeSH Terms: conditions — Obesity; Body Weight | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control without Metformin (No Intervention): Conventional management of obesity including basic instructions on diet and physical activity
- Control with Metformin (Experimental): Conventional management of obesity including basic instructions on diet and physical activity plus Metformin treatment
  Interventions: Drug: Metformin
- Intervention with Metformin (Experimental): Intensive physical activity course twice per week and monthly diet control by dietitian plus Metformin treatment.
  Interventions: Drug: Metformin
- Intervention without Metformin (No Intervention): Intensive physical activity course twice per week and monthly diet control by dietitian

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg BID for 12 months
  Other Names: Metforal
  Arms: Control with Metformin; Intervention with Metformin

SUMMARY:
The investigators hypothesize that Metformin decreases weight, normalizes lipid profile and increases insulin sensitivity; the study team hope to get better effect of weight decrease and metabolic processes repair in the intensive treatment group with intervention of physical activity, diet correction and Metformin use.

DETAILED DESCRIPTION:
During the first visit, study participants would follow the clinical investigation (anthropometry, physical examination, blood tests (hormonal and biochemical state), bioimpedance, ultrasound evaluation) and be attributed into 4 groups (matched for age, gender, pubertal stage and BMI), 100 subjects in each group.

1. st group - control: during the first visit patients get standardized information on healthy lifestyle, diet and exercise. Next visit (control) will be scheduled for the clinical and laboratory evaluation after 12 months of intervention.
2. nd group - intensive diet and physical activity group: Children will be seen

   1. by a dietician once a month for diet re-evaluation;
   2. physical therapist, who will give physical activity course twice a week (1 h each).
   3. pediatric endocrinologist every 3 months. Clinical and laboratory evaluation after 12 months of intervention.
3. rd group - intensive diet and physical activity group plus insulin sensitization: Metformin will be prescribed for this group of study children in the doses of 1000 mg/day Children will be seen by

   1. a dietician once a month for diet re-evaluation;
   2. physical therapist, who will give physical activity course twice a week (1 h each);
   3. pediatric endocrinologist every 3 month. Clinical and laboratory evaluation after 12 months of intervention.
4. th group- insulin sensitization without intensive diet and physical activity. Metformin will be prescribed in the doses of 1000 mg/day after standardized information on healthy lifestyle, diet and exercise during the first visit only. This group of children will be seen by pediatric endocrinologist every 3 months.

Intervention duration - 12 months. In the case of Metformin intolerance, children will continue the study in 2nd group.

Clinical and laboratory evaluation after 12 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17 yrs;
* Weight > 85th percentile for age and gender (by IOTF);
* Living in Kaunas and its region;
* No obvious chronic diseases;
* Not on steroid or other long-term treatment;
* Informed consent of the patient and parents (official caregivers);

Exclusion Criteria:

* Age less than 10 or above 17 yrs;
* Diagnosis of type 1 diabetes;
* Chronic illness that may affect physical activity and metabolic profile;
* Insulin treatment;
* Steroid treatment;
* Planning to move from Kaunas or its region in the period of 1 year;
* Protocol refused by the patient or his parents;

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Body mass index changes | 12 months
  decrease in body mass index

SECONDARY OUTCOMES:
Glucose homeostasis | 12 month
  Insulin sensitivity increase, homeostasis model assessment (HOMA-IR) decrease, insulin and glucose concentrations normalisation
Lipid profile | 12 months
  Lipid profile normalisation
Metabolic syndrome | 12 months
  Metabolic syndrome prevalence and risks decrease
Hepatosteatosis | 12 months
  Hepatosteatosis prevalence decrease and liver function improvement, hepatic enzymes normalisation
Polycystic ovary syndrome (PCOS) and hyperandrogenism in females | 12 months
  PCOS clinical symptoms regression, menstrual cycle normalisation, hirsutism, androgens levels decreasing and estrogen, sex hormone-binding globulin (SHBG) levels increasing

OTHER OUTCOMES:
safety | 12 months
  how many patients will have adverse events and withdraw the Metformin due to their intolerance or clinical / biochemical relapse

CONTACTS AND LOCATIONS:
Overall Officials: Rasa Verkauskiene, Professor, Study Chair — Lithuanian University of Health Sciences Hospital, Endocrinology Unit
Locations (1):
- Rasa Verkauskiene, Kaunas, Eiveniu Str. 2, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided
Study results are in progress with statistical analysis